CLINICAL TRIAL: NCT02348372
Title: A Phase I, Randomized, Single-Blind, Placebo-Controlled, Dose-Escalation (Part 1), Fixed Sequence and Open-Label (Part 2), Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Single Oral Doses of GSK1278863A in Healthy Subjects
Brief Title: Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Single Oral Doses of GSK1278863A in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 115385
Record Dates: First submitted 2012-04-05; First posted 2015-01-28 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Anaemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant

ARMS (5):
- GSK1278863A Placebo (Placebo Comparator): 5, 25 and 100 mg matched
  Interventions: Drug: GSK1278863A Placebo; Drug: GSK1278863A
- GSK1278863A 10mg (Experimental): A round, biconvex, white film coated tablet
  Interventions: Drug: GSK1278863A Placebo; Drug: GSK1278863A
- GSK1278863A 25mg (Experimental): A round, biconvex, white film coated tablet
  Interventions: Drug: GSK1278863A
- GSK1278863A 50mg (Experimental): A round, biconvex, white film coated tablet
  Interventions: Drug: GSK1278863A
- GSK1278863A 100mg (Experimental): A round, biconvex, white film coated tablet
  Interventions: Drug: GSK1278863A

INTERVENTIONS:
Drug: GSK1278863A Placebo — Matching size, shape and color
  Arms: GSK1278863A 10mg; GSK1278863A Placebo
Drug: GSK1278863A — A round, biconvex, white film coated tablet

SUMMARY:
GSK1278863A is a novel small molecule agent, which stimulates erythropoiesis through inhibition of hypoxia-inducible factor (HIF)-prolyl hydroxylases (EGLNs). This compound is being developed for the treatment of anemia. This study, PHI115385, will be the first administration of GSK1278863A to Japanese subjects to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single oral doses in healthy Japanese adult subjects. Healthy Caucasian adult subjects will be included in order to compare pharmacokinetics of GSK1278863A and its metabolite(s), and pharmacodynamics of GSK1278863A.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin >1.5xULN.
* Healthy Male or female between 20 and 65 years of age inclusive, at the time of signing the informed consent.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods.
* Body weight > 50 kg and BMI within the range 18.5 - 29.0 kg/m2 (inclusive).
* Capable of giving written informed consent.
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* Japanese defined being born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese. Japanese subjects should be also have lived outside Japan for less than 10 years.
* Caucasian, defined as an individual having four grandparents who are all descendents of the original peoples of Europe.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines
* A hemoglobin value at Screening is of: Healthy male subjects or post-menopausal females: > 16.5 g/dL, Healthy female (non-childbearing potential) subjects: > 15.5 g/dL
* The values of hematological parameters at screening are: MCV: outside the reference range and deemed clinically significant by the investigator and GSK Medical Monitor.
* The values of the following tests at Screening, for healthy subjects are: TIBC: outside the reference range of the population being studied, Serum iron: outside the reference range of the population being studied, Serum ferritin: outside the reference range of the population being studied
* A value at screening is greater than the upper limit of reference range for the following clinical laboratory parameters: AST, ALT, direct bilirubin.
* Clinically significant abnormal CPK determined by the Investigator and GSK Medical Monitor.
* Calculated creatinine clearance: < 80 mL/min
* A positive test for HIV antibody
* History of drug abuse or dependence within 6 months of the study.
* History of regular alcohol consumption within 6 months of the study
* History or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. By exception, subject may take acetaminophen (<2 grams/day) up to 48 hours prior to the first dose of study drug.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinical research unit uses heparin to maintain intravenous cannula).
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, and/or hepatic function that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Examples of conditions that could interfere with normal gastrointestinal anatomy or motility include cholecystectomy, gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, or celiac sprue. Examples of conditions that could interfere with hepatic function include Gilberts syndrome.
* History of peptic ulcer disease or chronic rectal bleeding.
* History of malignancy. Non-melanoma skin cancer that has been definitely removed is allowed.
* Subjects with a baseline medical history of proliferative diabetic retinopathy, preproliferative diabetic retinopathy, or wet age-related macular degeneration (AMD).
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures, or lifestyle and/or dietary restrictions outlined in the protocol.
* Consumption of >3 servings per day of red wine, grapefruit (juice), blood orange (juice), star fruit, onions, kale, broccoli, green beans, or apples from 7 days prior to the first dose of investigational product, unless in the opinion of the Investigator and GSK Medical Monitor this will not interfere with the study procedures and compromise subject safety.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Subject is mentally or legally incapacitated.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-03-31 (Actual); Primary Completion 2011-06-03 (Actual); Study Completion 2011-06-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 96 hr
AUC(0-t), AUC(0-∞), Cmax, tmax and t½ of GSK1278863A | up to 96 hr
Changes from Baseline of Clinical laboratory tests | 0,2448 and 96 hr
  Platelet Count , RBC Indices, WBC Differential, RBC Count, WBC Count, Lymphocytes, Reticulocyte Count, Hemoglobin, Hematocritm, BUN, Ptassium, AST, Total and direct bilirubin, Creatinine, Chloride, ALT, Uric Acid, Glucose, Total CO2, GGT, Albumin, Sodium, Calcium, Alkaline phosphatase, Total Protein, CPK, Iron Ferritin, TIBC
Changes from Baseline of Vital signs | 0, 1,2,3,4,8 and 24hr
  systolic and diastolic blood pressure and pulse rate
Change from Baseline of 12-lead ECG | 0,4 and 8 hr

SECONDARY OUTCOMES:
Hemoglobin endpoints: Hemoglobin actual values, change from baseline, rate of rise/decline, maximum change from baseline, and maximum % change from baseline | up to 96 hr

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115385 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115385?search=study&search_terms=115385#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 115385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register